CLINICAL TRIAL: NCT02083146
Title: C1q/TNF-related Proteins in Coronary Artery Disease
Status: Terminated | Type: Observational
Why Stopped: Study subjects were not enrolled.
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: CAD(CTRP)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Newly-developed ELISA was used for measurement of CTRP.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with CAD: Acute coronary syndromoe (ACS) patients who were admitted to the coronary care unit.

SUMMARY:
Now, adipose tissue is established as an active endocrine organ that controls systemic energy homeostasis by secretion of adipokines. Recently, members of the C1q/tumor necrosis factor-related protein (CTRP) family have been reported to share structural homology with adiponectin. To date, 15 CTRP family members have been found that might play major roles in metabolism and inflammation. The investigators tried to clarify the relationship between CTRP family and coronary artery disease (CAD) in Korean men and women.

DETAILED DESCRIPTION:
Adipose tissue secretes various kinds of bioactive molecules termed adipokines which contribute to the development of obesity-related disorders including cardiovascular disease (CVD). Adiponectin is the insulin-sensitizing adipokine with anti-inflammatory and anti-atherogenic properties. Hypoadiponectinemia has been associated with an increased risk of coronary artery disease (CAD) in several though not all studies. Recently, a new family of secreted proteins, C1q/TNF-related protein (CTRP), was cloned on the basis of sequence homology with adiponectin. This family of adiponectin paralogs might have pivotal implications in energy homeostasis and obesity-related inflammation. Each CTRP family member has its own unique tissue expression profile and function in regulating glucose and/or fat metabolism. In the present study, we evaluated the role of CTRP in patients with CAD and investigated whether CTRP family is significantly associated with CAD prevalence after adjustment for well-known CAD risk factors.

ELIGIBILITY:
Inclusion Criteria:

* 20<age<80
* History of stable angina, unstable angina, or acute myocardial infarction

Exclusion Criteria:

* a history of diabetes
* stage 2 hypertension
* malignancy
* severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects with stable angina or a history of acute coronary syndrome who visited for a department of cardiology in Korea Univ. Guro hospital were enrolled using predefined inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
serum concentration of CTRP-1,3, or 9 in the subjects with/without CAD | at enrollment
  compare serum concentration of CTRP-1,3 or 9 between CAD patients and normal group

SECONDARY OUTCOMES:
The relationships of serum CTRPs/adiponectin levels with cardiometabolic risk profiles | at enrollment
  find the correlation of CTRPs and adiponection with cardiometabolic risk

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, M.D., Principal Investigator — medica7@gmail.com
Locations (1):
- Korea Univ. Guro Hospital, Seoul, South Korea